CLINICAL TRIAL: NCT03859037
Title: Effect of Umbilical Cord Milking on Transition of Preterm Babies During Resuscitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Atef Elbeltagy, Principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AinshamsU12345; Aaaaaa (Registry Identifier: Ahmed)
Record Dates: First submitted 2019-02-11; First posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Fetal Distress
MeSH Terms: conditions — Fetal Distress | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Intervention Model Description: Two groups,one will have umbilical cord milking and other will have immediate cord clamping ,two groups will put on warmer after birth and blood pressure,heart rate ,oxygen saturation will be assessed by monitor every 30 seconds up to 10 minutes
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Umbilical cord milking (Experimental): One group will have umbilical cord milking and will ba assessed for blood pressure,oxygen saturation and heart rate by monitor
  Interventions: Other: Umbilical cord milking
- Immediate cord clamping (Placebo Comparator): One group will have immediate cord clamping and will be assessed for bloob pressure,heart rate,oxygen saturation by monitor
  Interventions: Other: Umbilical cord milking

INTERVENTIONS:
Other: Umbilical cord milking — 100 babies will have squeezing of blood from umbilical cord towards baby
  Other Names: Immediate cord claming

SUMMARY:
Investigators will evaluate if milking of umbilical cord in preterm babies will improve transition during resuscitation or not

DETAILED DESCRIPTION:
Investigators will make milking for 100 preterm babies and placed them on warmer and assess heart rate,blood pressure,oxygen saturation,fio2,maximum pip,PEEP and 100 babies other without milking to see the difference between two groups.

ELIGIBILITY:
Inclusion Criteria:

* babies who need resuscitation
* Preterm babies with 28-34 weeks gestatinal age

Exclusion Criteria:

* preterm babies above 34 weeks gestational age, -- -
* refusal by mother or obestatracain, -- -babies with congenital anomalies

Ages: 28 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2019-03-30 (Estimated); Study Completion 2019-04-10 (Estimated)

PRIMARY OUTCOMES:
measure mean blood pressure | Changes of all data will be assessed every 30seconds for ten minutes
  Measure mean blood pressure in mmhg

SECONDARY OUTCOMES:
Measure heart rate | Heart rate will be assessed every 30 seconds for 10 minuets
  Measure heart rate in beat/minutes

IPD SHARING:
Plan to Share IPD: Undecided